CLINICAL TRIAL: NCT03354754
Title: A Randomized, Controlled, Evaluator-blinded, Multi-center Study to Evaluate LYS228 Pharmacokinetics, Clinical Response, Safety, and Tolerability in Patients With Complicated Intra-abdominal Infection
Brief Title: LYS228 PK, Clinical Response, Safety and Tolerability in Patients With Complicated Intra-abdominal Infection (cIAI)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was closed as part of the out-licensure of the drug to Boston Pharmaceuticals, which will continue further clinical development of LYS228/BOS-228
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CLYS228X2202
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Results first posted 2019-10-08 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Intra-abdominal Infections
Keywords: Intra-abdominal infection; LYS228; beta-lactam antibiotics; creatinine clearance; enterobacteriaceae
MeSH Terms: conditions — Intraabdominal Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blinded evaluator performed the safety and efficacy assessments
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LYS228 (Experimental): IV infusion every 6 hours for at least 5 days
  Interventions: Drug: LYS228
- Standard of care (Active Comparator): IV infusion of standard of care antibiotics for at least 5 days
  Interventions: Drug: Standard of care therapy

INTERVENTIONS:
Drug: LYS228 — LYS228 IV infusion every 6 hours
  Arms: LYS228
Drug: Standard of care therapy — IV infusion of standard of care antibiotics
  Arms: Standard of care

SUMMARY:
The purpose of the study was to evaluate whether LYS228 can be developed for the treatment of complicated intra-abdominal infections.

It was planned that LYS228 exposure across patients with varying renal function would be evaluated during the study to confirm that LYS228 concentrations are predicted to be adequate to treat the patient population. It was planned that the PK exposure of the initial 8 patients would be analyzed.

PK analysis was not conducted as per protocol the first analysis required 8 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 to 85 years of age with visual confirmation (presence of pus within the abdominal cavity) of an intra-abdominal infection associated with peritonitis including at least one inclusionary diagnosis during surgical intervention.

Exclusion Criteria

* Any of the excluded diagnoses: abdominal wall abscess, small bowel obstruction, traumatic bowel perforation undergoing surgery within 12 hours, perforation of gastroduodenal ulcer with surgery within 24 hours, an intra-abdominal process that is not likely caused by infection.
* Pre-operative treatment of any duration with non-study Drug systemic antibiotic therapy for peritonitis or abscess is not allowed unless certain criteria are met.
* Concomitant bacterial infection at time of enrollment requiring non-Study Drug antibiotics and that may interfere with the evaluation of clinical response to the study antibiotic.
* Known non-abdominal source of infection, including endocarditis, osteomyelitis, abscess, meningitis, or pneumonia diagnosed within 7 days prior to enrollment.
* Patient has an Acute Physiology and Chronic Health Evaluation II (APACHE II) score > 30 or is considered, in the judgement of the investigator, unlikely to survive 4 weeks (e.g. rapidly progressive terminal illness, including septic shock).
* Patients that meet sepsis criteria as defined by the quick sequential sepsis-related organ failure assessment (qSOFA).
* Women of child-bearing potential unless they are using highly effective methods of contraception during dosing and for 7 days after stopping study treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Somers Point, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dean CR, Barkan DT, Bermingham A, Blais J, Casey F, Casarez A, Colvin R, Fuller J, Jones AK, Li C, Lopez S, Metzger LE 4th, Mostafavi M, Prathapam R, Rasper D, Reck F, Ruzin A, Shaul J, Shen X, Simmons RL, Skewes-Cox P, Takeoka KT, Tamrakar P, Uehara T, Wei JR. Mode of Action of the Monobactam LYS228 and Mechanisms Decreasing In Vitro Susceptibility in Escherichia coli and Klebsiella pneumoniae. Antimicrob Agents Chemother. 2018 Sep 24;62(10):e01200-18. doi: 10.1128/AAC.01200-18. Print 2018 Oct. PMID 30061293
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=769

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 60 patients were planned to be randomized to LYS228 or a comparator (standard of care therapy preferably piperacillin/tazobactam) in a 2:1 ratio.
Period: Overall Study
Arm/Group | LYS228 | Standard of Care
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LYS228 | Standard of Care | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Median (Full Range); unit: years] | 63.5 [63 to 64] | 63 [63 to 63] | 63 [63 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success at Day 28
Description: Clinical success is defined as resolution, or substantial improvement (i.e. reduction of severity of all baseline signs and symptoms and worsening of none) of all or most baseline signs and symptoms of cIAI infection without the need for additional antibiotic therapy other than any oral antibiotics given to complete treatment at home following discontinuation of Study Drug and no drainage or surgical reintervention required 96 hours after the start of Study Drug.
Time Frame: Day 28
Population: All patients
Measure: Count of Participants; unit: Participants
Arm/Group | LYS228 | Standard of Care
Number analyzed (Participants) | 2 | 1
Participants | 2 | 0

2. Primary Outcome: Plasma Pharmacokinetics (PK) of LYS228: Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau (AUCtau)
Description: Calculated based on LYS228 concentration in blood at different time points following drug administration on Day 5
Time Frame: Day 5
Population: PK analysis for the 2 patients enrolled that received LYS228 was not conducted as per protocol the first analysis required 8 patients.
Arm/Group | LYS228 | Standard of Care
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Plasma Pharmacokinetics (PK) of LYS228: The Observed Maximum Plasma Concentration Following Drug Administration (Cmax)
Description: Calculated based on LYS228 concentration in blood at different time points following drug administration on Day 5
Time Frame: Day 5
Population: as for outcome 2
Arm/Group | LYS228 | Standard of Care
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Plasma Pharmacokinetics (PK) of LYS228: The Time to Reach the Maximum Concentration After Drug Administration (Tmax)
Description: Calculated based on LYS228 concentration in blood at different time points following drug administration on Day 5
Time Frame: Day 5
Population: as for outcome 2
Arm/Group | LYS228 | Standard of Care
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Plasma Pharmacokinetics (PK) of LYS228: The Systemic (or Total Body) Clearance From Plasma Following Intravenous Administration (CL)
Description: Calculated based on LYS228 concentration in blood at different time points following drug administration on Day 5
Time Frame: Day 5
Population: as for outcome 2
Arm/Group | LYS228 | Standard of Care
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Plasma Pharmacokinetics (PK) of LYS228: The Volume of Distribution at Steady State Following Intravenous Administration (Vss)
Description: Calculated based on LYS228 concentration in blood at different time points following drug administration on Day 5
Time Frame: Day 5
Population: as for outcome 2
Arm/Group | LYS228 | Standard of Care
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Plasma Pharmacokinetics (PK) of LYS228: The Terminal Elimination Half-life (T1/2)
Description: Calculated based on LYS228 concentration in blood at different time points following drug administration on Day 5
Time Frame: Day 5
Population: as for outcome 2
Arm/Group | LYS228 | Standard of Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Patients With Adverse Events
Description: Number of patients with at least one Adverse Event
Time Frame: Daily
Population: All patients
Measure: Count of Participants; unit: Participants
Arm/Group | LYS228 | Standard of Care
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

9. Secondary Outcome: Microbiological Response at Day 28
Description: Microbiologic success at 28 days after randomization determined by microbial growth in culture from the intra-abdominal focus of infection when available or presumed eradication based on clinical success
Time Frame: Day 28
Population: All patients with a microbiological response assessment
Measure: Count of Participants; unit: Participants
Arm/Group | LYS228 | Standard of Care
Number analyzed (Participants) | 2 | 0
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until day 28.
Arm/Group | LYS228 | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LYS228 (N=2) | Standard of Care (N=1)
Appendicitis perforated (Infections and infestations) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LYS228 (N=2) | Standard of Care (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT03354754/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT03354754/SAP_001.pdf